CLINICAL TRIAL: NCT01520779
Title: Risk Factors for Recurrence of Hepatocellular Carcinoma After Radiofrequency Ablation
Brief Title: Recurrence of Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: HCC recurrence after RFA
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular cacinoma; Radiofrequancy ablation; Intrahepatic recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with recurrence: Hepatocellular carcinoma patients with intra-hepatic or distant recurrence of hepatocellular carcinoma within 1 year after radiofrequency ablation
- Patients with no recurrence: Hepatocellular carcinoma with no intra-hepatic or distant recurrence of hepatocellular carcinoma within 1 year after radiofrequency ablation

SUMMARY:
analysis of the risk factors of intra-hepatic distant recurrence (IDR) of hepatocellular carcinoma within 1 year after radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Proved diagnosis of HCC according to AASLD practice guidelines (Bruix and Sherman, 2005).
2. Patients underwent RFA for HCC with BCLC (The Barcelona-Clinic- Liver-Cancer staging system) stage A (Bruix and Sherman, 2005) with no eligibility or ability to do transplantation or resection.
3. Patients should be followed-up for more than 12 months to exclude early recurrence i.e. recurrence within 1 year.
4. Patients with INR < 1.5 or prothrombin concentration > 50%.
5. Platelet count > 50000 cell/mm3.

Exclusion Criteria:

1. Presence of extra-hepatic metastasis or gross vascular invasion.
2. Child class C patients.
3. Follow up period of less than 12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma (HCC) who underwent radiofrequency ablation (RFA) from 1/2006 till 12/2010in Tropical medicine department and hepatocellular carcinoma clinic, Ain Shams university
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of hepatocellular carcinoma | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Cairo, Egypt